CLINICAL TRIAL: NCT00548210
Title: Dermatix; A Randomized Controlled Trial Measuring Effectivity of Dermatix in Promoting Scar Maturation of Hypertrophic Scars.
Brief Title: Effectivity of Dermatix in Promoting Scar Maturation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association of Dutch Burn Centres (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Other Study IDs: DERMO0501
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Hypertrophic Scars
Keywords: Hypertrophy; scarring; scar treatment; silicone
MeSH Terms: conditions — Cicatrix, Hypertrophic; Hypertrophy; Cicatrix

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this research is to demonstrate effectivity of Dermatix in promoting maturation of the scar, versus a control region that will be treated with an indifferent cream.

DETAILED DESCRIPTION:
The healing of deep thermal injuries is always associated with scarring. The healing process can lead to the formation of large scar bundles (e.g. hypertrophic scars). The scars can be discomforting, disfiguring and restrict motion if situated over or near joints. Evidence for effectivity of treatment for reduction of hypertrophic scars or the prevention of them is limited.

Different treatments are used such as intralesional injected steroids, topically used oily creams, silicone sheets or occlusive dressings. Compression garments are also frequently used. There is some evidence as to the effectivity of silicone sheets for recuction of hypertrophic scarring, however, these sheets cannot be used easily on all anatomical locations.

Valeant Pharmaceuticals International has developed a silicone based scar remodelling gel, Dermatix®, which has been empirically shown by others to have potential to reduce hypertrophic scars.

Primary objectives are to demonstrate effectivity of Dermatix in promoting maturation of the scar, versus a control region that will be treated with an indifferent cream.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hypertrophic scarring and/or ropes, stable for at least 3 months before inclusion.
2. Written informed consent
3. Scar size enabling the definition of two distinct scar areas, with similar scar characteristics at inclusion, preferably symmetric scars.
4. Patients of 18 years or older

Exclusion criteria:

1. Known sensitivity for occlusive dressings or silicone containing products
2. Any patient condition that may influence the compliance of the treatment negatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Middelkoop, PhD, Study Director — Association of Dutch Burn Centres
Locations (1):
- Association of Dutch Burn Centres, Beverwijk, North Holland, Netherlands